CLINICAL TRIAL: NCT02796300
Title: Comparison of the Palindrome vs. BioFlo DuraMax Hemodialysis Catheters: A Prospective Randomized Trial
Brief Title: Study to Compare Palindrome vs. BioFlo DuraMax Dialysis Catheters
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor decided to terminate the study.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Principal Investigator, Edward Wolfgang Lee, MD, MD, PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLA Bioflo 2016
Record Dates: First submitted 2016-05-24; First posted 2016-06-10 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Chronic Kidney Disease
Keywords: bioflo; Duramax catheter; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bioflo Goup (Active Comparator): This group will have dialysis using the Bioflo catheter.
  Interventions: Device: Bioflo Dialysis Catheter
- Palindrome Group (Active Comparator): This group will have dialysis using the Palindrome catheter.
  Interventions: Device: Palindrome Dialysis Catheter

INTERVENTIONS:
Device: Bioflo Dialysis Catheter — The catheter placement procedure will be performed in the interventional radiology suite. The catheter will be inserted subcutaneously through incision in the chest through the tract.
  Arms: Bioflo Goup
Device: Palindrome Dialysis Catheter — The catheter placement procedure will be performed in the interventional radiology suite. The catheter will be inserted subcutaneously through incision in the chest through the tract.
  Arms: Palindrome Group

SUMMARY:
Numerous catheter designs have been studied to increase efficacy and minimize complications of catheter hemodialysis. Major complications of catheters include thrombosis, central venous stenosis, infection, and dialysis inadequacy. Thrombosis must be avoided if possible because using too many catheters may exhaust all of the catheter insertion sites on the body, as well as increase the risk of infection. This prospective study compares the complications and general outcomes of patients who receive hemodialysis using the mainstream Palindrome catheter versus the newer BioFlo DuraMax catheter.

This study will examine outcomes of patients who receive hemodialysis using either the Palindrome catheter or the BioFlo catheter. Patients will be observed and outcomes will be recorded for three to six months. Outcomes will be analyzed and compared to draw conclusions on which catheter produces less catheter thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 - 65 years of age;
2. First de novo dialysis catheter placement or second catheter exchange, no more than 3 replacements on a same site
3. Requiring at least 3 months dialysis catheter usage
4. No clinical or radiographic evidence of superior vena cava (SVC) narrowing
5. Patent right internal or external jugular vein
6. Willing to provide the dialysis center information for F/U
7. No known diagnosis of hypercoagulopathy

Exclusion Criteria:

1. Short term catheter usage plan (< 1 months)
2. No right jugular venous access
3. Catheter use for bone marrow transplant or plasmapheresis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lee, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 01/2017 to 12/2018 Location = UCLA Santa Monica Hospital
Pre-assignment Details: No significant events occurred in this study prior to assignment to a group
Period: Overall Study
Arm/Group | Bioflo Goup | Palindrome Group
Started | 10 | 22
Completed | 10 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bioflo Goup | Palindrome Group | Total
Number analyzed (Participants) | 10 | 22 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 2 | 12 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (14.7) | 61.2 (18.6) | 57.8 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 15 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 22 | 32

OUTCOME MEASURES:

1. Primary Outcome: Catheter Thrombosis Rate of Bioflo Catheters vs. Palindrome Catheters.
Description: A comparison of the number of tPA used as an indicator of thrombosed catheter per month between two groups
Time Frame: 1 month
Measure: Mean (Standard Error); unit: catheter thrombosis per month
Arm/Group | Bioflo Goup | Palindrome Group
Number analyzed (Participants) | 10 | 22
catheter thrombosis per month | 4.3 (0.56) | 7.27 (0.49)

2. Secondary Outcome: Catheter Thrombosis Rate of Bioflo Catheters vs. Palindrome Catheters.
Description: A comparison of the number of tPA used as an indicator of thrombosed catheter per month between two groups in three month follow-up
Time Frame: 3 months
Population: Two patients in the Palindrome group were not included in this outcome measure analysis. One patient received the kidney transplant during the 3 month follow-up and the second patient died during the 3 month follow-up
Measure: Mean (Standard Error); unit: catheter thrombosis per 3 months
Arm/Group | Bioflo Goup | Palindrome Group
Number analyzed (Participants) | 10 | 20
catheter thrombosis per 3 months | 8.6 (0.81) | 12.4 (1.07)

3. Secondary Outcome: Catheter Thrombosis Rate of Bioflo Catheters vs. Palindrome Catheters.
Description: If necessary, we will monitor the catheter thrombosis rate of Bioflo catheters vs. Palindrome catheters.
Time Frame: 6 months
Population: 6 month data were not collected due to a stopping rule invoked after the 3-month data were analyzed
Arm/Group | Bioflo Goup | Palindrome Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cost Analysis
Description: To perform a cost-analysis and economic burden of using Bioflo catheters compared to Palindrome catheters due to catheter thrombosis and exchange.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: US Dollar
Arm/Group | Bioflo Goup | Palindrome Group
Number analyzed (Participants) | 10 | 20
US Dollar | 60200 (5638.75) | 78909 (8716.53)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Bioflo Goup | Palindrome Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 3/22
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 0/10 | 0/22

LIMITATIONS AND CAVEATS:
An early termination occurred due to the decision made by the sponsor and PI. This led to smaller numbers of subjects analyzed than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT02796300/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02796300/ICF_001.pdf